CLINICAL TRIAL: NCT03694457
Title: Comparison Between Anterior Approach (Deltopectoral) and Lateral Approach (Deltoid Splitting) in Shoulder Reverse Arthroplasty for Proximal Humerus Fracture
Acronym: DELTOSUPEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-410; 2018-A02113-52 (Other: 2018-A02113-52)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Humeral Fracture; Aged Patient; Reversed Total Shoulder Arthroplasty; Surgical Approach
Keywords: Prospective; Randomized study; Proximal humerus fracture; Surgical treatment
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deltopectoral approach (Active Comparator): the patients are treated with deltopectoral approach surgery
  Interventions: Procedure: Reversed total shoulder arthroplasty
- lateral approach (Other): the patients are treated with a lateral approach surgery
  Interventions: Procedure: lateral approach

INTERVENTIONS:
Procedure: Reversed total shoulder arthroplasty — Replacement of the proximal humeral head by a reversed prosthesis through an anterior approach
  Arms: deltopectoral approach
Procedure: lateral approach — Replacement of the proximal humeral head by a reversed prosthesis through a lateral approach
  Arms: lateral approach

SUMMARY:
The aim of the study consists in comparing two surgical approaches (deltopectoral versus lateral deltoid splitting) in the treatment of proximal humerus fractures treated with a reversed total shoulder arthroplasty The assessment will focus on clinical (clinical scores, efficacy, safety…) and radiological results, between these two types of surgical approaches by using a prospective, randomized analysis.

DETAILED DESCRIPTION:
The 2 main surgical approaches in total shoulder arthroplasty (TSA) are the anterior approach (deltopectoral) and the lateral one (deltoid splitting) (18).

Their advantages and drawbacks have not been clearly evaluated in proximal humerus fracture treated with an arthroplasty.

The goal of the study is to compare the results between patients (older than 65yo) presenting a proximal humerus fracture treated with a reversed shoulder arthroplasty performed through an anterior approach or a lateral one.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 65yo with a proximal humerus fracture (Neer 3-4 and 2 dislcated)
* Patient registered to the national health system
* Patient able to understand information about the protocol and answer to questionnaire

Exclusion Criteria:

* Non-displaced fracture or no need of surgical treatment.
* Existing bone disease
* Infection
* Neurological deficit (axillary nerve)
* Multi-injured patients
* Patient no able to fulfill the questionnaire
* Patient refuses the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Constant Murley Score | 12 months
  Constant Murley Score it a clinical method of functional assessment of the shoulder. The score varies between 0 and 100, more the value is better brought up is the score

SECONDARY OUTCOMES:
Quick dash score | 3, 6 and 12 months
  the Quick Dash score is a functional assessment of the shoulder. The score varies between 0 and 100, more the value is better brought up is the score
SF12 score | 3, 6 and 12 months
  The SF12 score is a quality of life assessment. The score varies between 0 and 100, more the value is better brought up is the score
Alder score | 3, 6 and 12 months
  Assessment of external rotation of the shoulder. The score varies between 0 and 100, more the value is better brought up is the score
The Simple Shoulder Test (SST) | 3, 6 and 12 months
  The Simple Shoulder Test is functional assessment of the shoulder. The score varies between 0 and 100, more the value is better brought up is the score
WOOS (The Western Ontario Osteosarthritis ) | 3, 6 and 12 months
  The Western Ontario Osteosarthritis of the shoulder index is a quality of life measurement tool for osteoarthritis of the shoulder. The score varies between 0 and 100, more the value is better brought up is the score
intensity of pain | pre op, 3, 6 and 12 months
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
Radiologic evaluation | pre op, 3, 6 and 12 months
  Radiologic evaluation
Complications | pre op, 3, 6 and 12 months
  list of the complications

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume VILLATTE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196